CLINICAL TRIAL: NCT04838145
Title: The Diabetes Virus Detection and Intervention Trial
Acronym: DiViDInt
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Krogvold, Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-003350-41
Record Dates: First submitted 2019-01-04; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Type1 Diabetes Mellitus; Enterovirus
Keywords: Type 1 diabetes; Children; Enterovirus; Recent onset
MeSH Terms: conditions — Enterovirus Infections; Diabetes Mellitus, Type 1 | interventions — Ribavirin; pleconaril

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo controlled, prospective, randomized trial examining the effect of antiviral treatment given for 6months on residual insulin secretion
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Active Comparator): Pleconaril: 5 mg/kg x2 times a day for 26 weeks up to 40 kg. Max dose 300mg x2. Ribavirin:15 (7.5) mg/kg/day divided in two doses daily for 26 weeks: Max dose 1000mg/24h if body weight<75kg and 1200mg if body weight>75kg.
  Interventions: Drug: Ribavirin + Pleconaril
- Placebo (Placebo Comparator): Receives placebo, on a double blind basis
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Ribavirin + Pleconaril — Randomized to treatment with study drugs (ribavirin and pleconaril)
  Arms: Active treatment
Drug: Placebos — Randomized to treatment with placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled study in 96 children and adolescents age 6-15 newly diagnosed with type 1 diabetes to describe the influence of antiviral treatment (Pleconaril and Ribavirin) on progression of disease and residual insulin secretion.

DETAILED DESCRIPTION:
If antiviral treatment is efficient in halting the disease progression, it will be to great benefit for the participating patients. Maintenance or even an increase in beta cell mass due to regeneration will lead to improved endogenous insulin production and give a milder course of the disease with improved glycemic control. This will in a substantial way improve the long-term prognosis with less severe long term vascular complications.Some patients may have close to complete remission and be able to stop insulin treatment. If antiviral treatment is effective, it would add proof to the concept that type 1 diabetes in its origin is a viral disease. This would be an important milestone in medical research and a breakthrough in the understanding of the etiopathogenesis of autoimmune diseases. It may promote the development of vaccines to prevent the disease. T1D seems more aggressive in children than in adults, and the beta cell function decline rapidly compared to adults. As a consequence, the effect of antiviral treatment will potentially be more significant in children than in adults. Children have higher HbA1c which increases the risk of complications. Thus, T1D is a more aggressive disease in children than in adults and hence it's important to do this study in children. Pharmaceuticals are usually studied in different age intervals, commonly 1-6 years, 6-12 years and 12-15 years. For safety reasons and simplicity, the investigators want to start with the two older groups. The investigators will treat the participants with two antiviral medications (Pleconaril and ribavirin) or placebo in a double blind, randomized, placebo controlled, parallel group study. Pleconaril has previously been given in doses of 5-10mg/kg x 2-3 in clinical trials in children, thus achieving serum levels high enough for killing the majority of the viruses. The investigators have, due to the long treatment period, reduced the doses to 5 mg/kg x 2. Ribavirin will be given in dosages according to Summariy of product characteristics (SmPC). The investigators have chosen to administer Investigational Medicinal Product (IMPs) as an oral solution as this will make it easier to give the medication according to weight.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed type 1 Diabetes (E10.9). First injection of insulin maximum three weeks prior to inclusion.
2. Must be willing and capable of taking the study drugs and meet for tests and follow up as described.
3. Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to International Conference on Harmonization Good Clinical Practice (ICH GCP), and national/local regulations.
4. Aged 6.00-15.99 years at inclusion

Exclusion Criteria:

1. Treatment with any oral or injected anti-diabetic medications other than insulin.
2. A history of haemolytic anaemia or significantly abnormal haematology results at screening.
3. History of severe cardiac disease previous six months.
4. Impaired renal function
5. Patients taking ethinyl estradiol
6. Participation in other clinical trials with a new chemical entity within the previous 3 months.
7. Inability or unwillingness to comply with the provisions of this protocol
8. Females who are lactating or pregnant.
9. Males or females (after menarche) not willing to use highly effective contraception (progesterone-only hormonal anticonception with inhibition of ovulation or sexual abstinence) and barrier contraception (condoms), if sexually active during the treatment period and in the following 7 months
10. Presence of serious disease or condition, which in the opinion of the investigator makes the patient non-eligible for the study.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Insulin secretion | 12 months
  Change in mean residual insulin secretion in the Insulin tolerance test (ITT)-population measured by Mixed Meal Tolerance Test (MMTT) stimulated C-peptide two-hour area under the curve profile from visit 1 to12 months after initiation of study treatment.

SECONDARY OUTCOMES:
Insulin secretion | 3 months
  Change in mean residual insulin secretion in the ITT-population measured by Mixed Meal Tolerance Test (MMTT) stimulated C-peptide two-hour area under the curve profile from visit 1 to 3 months after initiation of study treatment.
Insulin secretion | 6 months
  Change in mean residual insulin secretion in the ITT-population measured by Mixed Meal Tolerance Test (MMTT) stimulated C-peptide two-hour area under the curve profile from visit 1 to 6 months after initiation of study treatment.
Insulin secretion | 24 months
  Change in mean residual insulin secretion in the ITT-population measured by Mixed Meal Tolerance Test (MMTT) stimulated C-peptide two-hour area under the curve profile from visit 1 to 24 months after initiation of study treatment.
Insulin secretion | 36 months
  Change in mean residual insulin secretion in the ITT-population measured by Mixed Meal Tolerance Test (MMTT) stimulated C-peptide two-hour area under the curve profile from visit 1 to 36 months after initiation of study treatment.
Stimulated c-peptide | 36 months
  Proportion of patients with peak residual insulin secretion measured by MMTT: stimulated C-peptide >0.2 pmol/L
C-peptide filter paper | 36 months
  Fasting and meal stimulated C-peptide from blood sampled on filter paper at home at 4 weekly intervals throughout the study period
Insulin dose | 36 months
  Mean Insulin dosage per kilo bodyweight per 24 hours
HbA1c | 36 months
  HbA1c at every control
Hypoglycemic events | 36 months
  Number of severe hypoglycaemic events and less severe events requiring assistance from others with blood glucose values ≤ 3.9 mmol/L will be registered at each control
Insulin-dose-adjusted HbA1c (IDAA1c) | 36 months
  HbA1c adjusted to insulin dose
Proinsulin/c-peptide ratio in serum | 36 months
  Proinsulin/c-peptide ratio in serum as a measure of beta cell stress
Presence of enterovirus | 36 months
  Presence of enterovirus and rhinovirus and/or neutralizing antibodies against those viruses in nose, blood, saliva and stool

CONTACTS AND LOCATIONS:
Overall Officials: Knut Dahl-Jørgensen, MD, PhD, Principal Investigator — Professor
Locations (1):
- Pediatric department, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
The data and material collected from the placebo-group will be shared with the "Innodia" consortium